CLINICAL TRIAL: NCT07218289
Title: Green Light Therapy to Reduce Pain and Promote Wellness After Surgery: A Randomized Controlled Trial in Adult Post-Operative Patients
Brief Title: Green Light for Post-Operative Wellness
Acronym: GLOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecca E Kotcher, MD (Other)
Responsible Party: Sponsor-Investigator, Rebecca E Kotcher, MD, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25080068
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Surgery
Keywords: light therapy; post-operative pain; depression; anxiety; post-operative recovery
MeSH Terms: conditions — Pain, Postoperative; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Bright Green Light Exposure Arm (Experimental): Subjects randomized to this group will be exposed to bright green light via the Day Light Classic Plus light therapy lamp fitted with an appropriate color filter. The light will be administered for 4 hours daily for up to three days post-operatively while the subject is in the hospital.
  Interventions: Device: Bright Green Light Therapy
- Dim White Light Exposure Arm (Active Comparator): Subjects randomized to this group will be exposed to dim white light via the Day Light Classic Plus light therapy lamp fitted with an appropriate color filter. The light will be administered for 4 hours daily for up to three days post-operatively while the subject is in the hospital.
  Interventions: Device: Dim White Light Therapy

INTERVENTIONS:
Device: Bright Green Light Therapy — Day Light Classic Plus light therapy lamp with filter to yield bright green light.
  Arms: Bright Green Light Exposure Arm
Device: Dim White Light Therapy — Day Light Classic Plus light therapy lamp with filter to yield dim white light.
  Arms: Dim White Light Exposure Arm

SUMMARY:
This is an unblinded, parallel group randomized controlled trial to evaluate bright green light as an adjunct therapy after surgery at UPMC Shadyside. The primary outcome measure will be pain intensity with secondary outcome measures including opioid requirements, sleep quality, mood, and overall post-operative recovery. Specific aims/hypotheses for this study are as follows:

Aim 1: To assess bright green light therapy's potential as a complementary post-operative analgesic strategy in patients recovering from surgery Hypothesis 1: Participants exposed to bright green light, in comparison to dim white (ambient) light, will have improved postoperative pain scores and lower opioid use.

Aim 2: To examine the impact of bright green light therapy on patient-centered measures of post-operative recovery that may be related to improved circadian function.

Hypothesis 2: Participants exposed to bright green light, in comparison to dim white (ambient) light, will have improved quality of post-operative recovery, enhanced sleep, and reduced anxiety and depression.

DETAILED DESCRIPTION:
This research study is being done to evaluate the use of light therapy following surgery at UPMC Shadyside Hospital (Pittsburgh, PA). Light therapy after surgery may reduce pain and pain medication requirements, and it may improve sleep, mood, and overall post-surgery recovery. The proposed study design of a randomized controlled trial investigates the use of bright green light therapy for post-operative pain management and wellness.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Planned to undergo laparoscopic or robotic surgery at UPMC Shadyside Hospital
* Anticipated post-operative length of stay >/= 48 hours
* Able to speak and read English fluently, with the capacity to provide informed consent and complete the associated surveys independently

Exclusion Criteria:

* Pregnancy
* History of significant ocular issues/dysfunction (†‡ ) (e.g., glaucoma, ocular trauma, macular degeneration, cataracts) that would interfere with the ocular mechanism of action
* History of significant neurological disease (‡) (e.g., traumatic brain injury, stroke, neurodegenerative disease) that would compromise the reliability of pain screening and/or interfere with the central mechanism of action
* History of bipolar disorder or schizophrenia, which could increase the risk of an adverse reaction to light exposure (i.e., acute mania)
* History of splenectomy, which would interfere with the mechanism of action

  * Ocular issues corrected with contact lenses or spectacle corrective eyeglasses will NOT be considered a criterion for exclusion ‡Unclear cases will be at the discretion of the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incisional Pain Intensity with Movement | Post-Operative Day 2
  Incisional pain with movement (after coughing) will be reported using a Numerical Rating Scale (NRS), scored from 0 to10, with 0 indicates "no pain" and 10 indicates "the worst pain imaginable". Post-intervention NRS on Post-Operative Day 2 will be compared between study arms as the primary outcome.

SECONDARY OUTCOMES:
Incisional Pain Intensity at Rest | Post-Operative Day 2
  Incisional pain at rest will be reported using a Numerical Rating Scale (NRS), scored from 0 to10, where 0 indicates "no pain" and 10 indicates "the worst pain imaginable". Post-intervention NRS on Post-Operative Day 2 will be compared between study arms as a secondary outcome.
Oral Morphine Equivalents (OME) | Post-Operative Day 1, and Post-Operative Day 2
  Total Opioid use will be obtained from the electronic medical record. Oral Morphine Equivalent (OME) use during the first 48-hours after surgery will be compared (on Post-Operative Days 1 and 2) between study arms.
Sleep Disturbance | Post-Operative Day 7
  Sleep disturbance will be assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disturbance 8-Item Short Form. Standardized T-scores (population mean = 50, standard deviation =10) will be compared between study arms as a secondary outcome. Higher scores will indicate higher levels of sleep disturbance.
Depression | Post-Operative Day 7
  Depression will be measured using the PROMIS (Patient-Reported Outcomes Measurement Information System) Depression 8-Item Short Form. Minimum score of 8, and Maximum score of 40. Higher scores will indicate higher levels of depression (worse outcome). Standardized T-scores (population mean = 50, standard deviation = 10) on post-operative Day 7 will be compared between study arms as a secondary outcome.
Anxiety | Post-Operative Day 7
  Anxiety will be assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) Anxiety 8-Item Short Form. Scores range from 8 to 40. Higher scores will indicate greater anxiety.
Overall quality of Post-Operative Recovery | on Post-Operative Day 2, and Post-Operative Day 7
  Overall recovery will be assessed using the Quality of Recovery-15 (QoR-15) questionnaire, scored from 0 to 150. Higher scores will indicate better recovery. QOR-15 will be compared between study arms as a secondary outcome on both of Post-Operative Day 2 and Post-Operative Day 7.
Hospital Length of Stay | Up to 30 Days Post-Operatively
  Hospital length of stay will be reported as the total of full days spent in an acute care hospital or emergency department within 30 days after surgery (0-30) and will be compared between study arms as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kotcher, MD, Principal Investigator — University of Pittsburgh, UPMC
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
In the future, the investigators may decide to share data with other investigators both within or outside of this institution. If this were to occur, the investigators would de-identify all of the information prior to sharing data in this way.